CLINICAL TRIAL: NCT07259395
Title: Prospective Validation of the SWEET Tool for Pre-diction of Preintervention ERCP Procedure Time.
Status: Recruiting | Type: Observational
Sponsor: Universitair Ziekenhuis Brussel (Other)
Responsible Party: Sponsor
Other Study IDs: TIME SWEET
Record Dates: First submitted 2025-11-14; First posted 2025-12-02 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-10

CONDITIONS: Endoscopic Retrograde Cholangio-Pancreatography
Keywords: SWEET tool; ERCP; Endoscopic Retrograde Cholangio-Pancreatography
MeSH Terms: interventions — Cholangiopancreatography, Endoscopic Retrograde

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- ERCP group
  Interventions: Procedure: ERCP

INTERVENTIONS:
Procedure: ERCP — Endoscopic retrograde cholangiopancreatography

SUMMARY:
Endoscopic retrograde cholangiopancreatography (ERCP) is a frequently performed procedure worldwide. The procedure combines endoscopy and X-ray imaging to diagnose and treat problems in the bile and pancreatic ducts, most commonly stones or strictures.

Until the recent publication of Waldthaler et al., there was little evidence about what patient- and procedure-related factors determine a priori the duration of an ERCP. Data from 74 248 ERCPs performed from 2010 to 2019 were extracted from the Swedish National Quality Registry (GallRiks) to identify variables predictive for ERCP time using linear regression analyses and root mean squared error (RMSE) as a loss function. Ten variables were combined to create an estimation tool for ERCP duration: the SWedish Estimation of ERCP Time (SWEET) tool. Having a predictive tool for estimating the procedure time of an invasive endoscopic procedure offers several valuable benefits across clinical, operational, and patient-centered domains: improved scheduling and resource allocation by optimized operating room and endos-copy suite scheduling, reduced delays and less overbooking or underutilization. It helps allocate the right number of staff (nurses, anesthesiologists) based on procedure complexity and minimizes unexpected extensions that lead to staff fatigue or overtime pay.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* First or redo-ERCP
* Intraductal endoscopy
* ERCPs performed by fellows under supervision

Exclusion Criteria:

* ERCPs in altered anatomy
* ERCPs combined with therapeutic EUS interventions

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients receiving an ERCP
Sampling Method: Non-Probability Sample
Enrollment: 363 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Accuracy of the time an ERCP procedure will take between the SWEET tool and the prediction of the endoscopist | From signing the ICF till end of the ERCP procedure.
  Accuracy of the SWEET (SWedish Estimation of ERCP Time) tool for predicting of ERCP preintervention procedure time compared to the prediction by the endoscopist.
Accuracy of the time the ERCP procedure will take between the SWEET tool and real time | From signing the ICF till end of the ERCP procedure.
  Accuracy of the SWEET (SWedish Estimation of ERCP Time) tool for predicting of ERCP preintervention procedure time compared to the measured real time.

SECONDARY OUTCOMES:
Predictors of Overestimation or Underestimation of ERCP Procedure Time (Difference in Minutes) | from signing the ICF till end of the ERCP procedure.
  Identify factors influencing over/underestimation of ERCP time by the performing endoscopist

CONTACTS AND LOCATIONS:
Locations (1):
- UZ Brussel, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No